CLINICAL TRIAL: NCT04260750
Title: ICBT for Depression - A Factorial Investigation of Kinds of Therapist Support and Self-/Expert-selected Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: LUNA
Record Dates: First submitted 2020-01-30; First posted 2020-02-07 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Depressive Disorder, Major; Depressive Symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Factor one: Regular therapist support by a therapist/On-demand guidance by a health care team (the participants themselves can choose to contact a physician, a nurse, a clinical psychologist, an IT-technician and/or the principal investigator of the study).
  Factor two: The content (the modules) is chosen by the participants themselves/The content is chosen by the therapist conducting the intake interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Expert-chosen content, regular guidance (Experimental): Content chosen by the therapist, weekly guidance by a therapist.
  Interventions: Behavioral: Internet-administered Cognitive behavioral therapy (ICBT)
- Expert-chosen content, on-demand guidance (Experimental): Content chosen by the therapist, guidance upon request from the health care team.
  Interventions: Behavioral: Internet-administered Cognitive behavioral therapy (ICBT)
- Participant-chosen content, regular guidance (Experimental): Content chosen by participants themselves, weekly guidance by a therapist.
  Interventions: Behavioral: Internet-administered Cognitive behavioral therapy (ICBT)
- Participant-chosen content, on-demand guidance (Experimental): Content chosen by participants themselves, guidance upon request from the health care team.
  Interventions: Behavioral: Internet-administered Cognitive behavioral therapy (ICBT)

INTERVENTIONS:
Behavioral: Internet-administered Cognitive behavioral therapy (ICBT) — The intervention consists of fifteen modules, each having a specific focus on a problem (e.g. comorbid worry alongside the depression) or containing a specific strategy or element (e.g. behavioral activation).
  The fifteen modules are:
  Introduction/Psychoeducation about depression, Behavioral activation 1, Behavioral activation 2, Cognitive restructuring, Acceptance, Psychoeducation about emotions, Anxiety and exposure, Comorbid social anxiety, Comorbid worrying and generalized anxiety, Comorbid panic disorder, Sleep problems, Perfectionism, Stress management, Relaxation, and Relapse prevention.
  The first and last module are assigned to all participants. The rest is picked either by the participants themselves or by the therapist conducting the intake interview.

SUMMARY:
The study is a factorial randomized controlled trial investigating the efficacy of difference versions of internet-administered cognitive behavioral therapy.

DETAILED DESCRIPTION:
The study is a 2 x 2 design. The first factor thought to be of relevance for the efficacy is the whether the content is selected by the participants themselves or by a therapist. The second factor consists of two levels: regular, continuous weekly support from a therapist or guidance on demand by a health care team consisting of a physician, a nurse, a clinical psychologist, an IT-technician and the principal investigator of the study.

ELIGIBILITY:
Inclusion Criteria:

* Current depressive symptoms equivalent to a score of at least 5 on Patient Health Questionnaire 9 and a minimum of 10 points on Becks Depression Inventory.
* 18 years or older.
* Adequate ability to understand and speak Swedish.
* Access to the internet and a smartphone/computer.

Exclusion Criteria:

* Other ongoing psychological treatment or counselling.
* Recent (within the past 3 months) changes in the dose of psychotropic medication.
* Prior diagnosis of psychosis, bipolar disorder, or substance dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Change on Becks Depression Inventory-II (BDI-II) | Baseline, after the intervention (after 11 weeks), 12 months after the end of intervention.
  Measure of depressive symptoms. Possible range for the total sum: 0 to 63 (created by summing up the score from each item). Clinical ranges for minimal, mild, moderate and severe major depressive disorder are considered to be 0-13, 13-19, 20-28, and 29-63 points.
Change on Patient Health Questionnaire (PHQ-9) | Baseline, during week 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10 of the intervention, post-intervention (after 11 weeks), 12 months after the end of intervention.
  Measure of depressive symptoms. Possible range for the total sum: 0 to 27 (created by summing up the score from each item). Clinical cut-offs for mild, moderate, moderately severe and severe major depressive disorder are considered to be 5, 10, 15, and 20 points.

SECONDARY OUTCOMES:
Change on Generalised Anxiety Disorder 7-item scale (GAD-7) | Baseline, after the intervention (after 11 weeks), 12 months after the end of intervention.
  Measure of symptoms of generalised anxiety disorder (GAD). Seven items, the score is interpreted by summing up the score from each individual item. Higher scores indicate more severe problems with worry and generalised anxiety. The total sum ranges from 0 to 21 with cut-offs of 5, 10, and 15 representing mild, moderate and severe generalised anxiety.
Change on Brunnsviken Brief Quality of Life Scale (BBQ) | Baseline, after the intervention (after 11 weeks), 12 months after the end of intervention.
  Measure of quality of life, total score ranging from 0 to 96 with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.
Change on Insomnia Severity Index (ISI) | Baseline, after the intervention (after 11 weeks), 12 months after the end of intervention.
  Measure of insomnia severity and symptoms of disordered sleep. The total score can range between 0 (no sleep problems) to 28 (severe sleep problems and insomnia). Norm score ranges include low likelihood of sleep problems (0 to 7 points), some sleep problems (8 to 14 points), moderate sleep problems (15 to 21 points), severe sleep problems (22 to 28 points).

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No